CLINICAL TRIAL: NCT02789124
Title: Diagnostic Value of Passive Leg Raise Induced Changes in Carotid Artery Flow Time to Predict Fluid Responsiveness in Critically Ill Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Mohamed Saad, PI, University of Louisville
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 14.0272
Record Dates: First submitted 2015-02-04; First posted 2016-06-02 (Estimated); Last update posted 2016-06-09 (Estimated); Status verified 2016-06

CONDITIONS: Fluid Responsiveness; Carotid Artery Flow Time; Passive Leg Raise
Keywords: fluid responsiveness; carotid artery flow time; passive leg raise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Carotid Artery Flow Time (Experimental): Patients with radial aline and flotrac vigileo will have carotid dopper measured for carotid flow time and a passive leg raise
  Interventions: Other: Carotid Doppler Measurement in response to passive leg raise

INTERVENTIONS:
Other: Carotid Doppler Measurement in response to passive leg raise — The investigators will measure Carotid Flow time in the semi-recumbent position, then lay the patient flat and do a passive leg raise. The investigators will then meausre Carotid Flow Time at 1 minute, 2 minutes, and 3 minutes. Patients who have 10 % increase in stroke volume on the Flotrac / Vigileo monitor will be considered fluid responders. The investigators will try to identify an optimum % increase of Carotid Flow Time that can predict fluid responsiveness.

SUMMARY:
Difficulties in the accurate assessment of intravascular volume in critically ill patients are frequently encountered. In addition to clinical evaluation, bedside echocardiographic measurements of fluid responsiveness can be technically difficult, especially in critically ill mechanically ventilated patients. The carotid artery is an easily accessible structure that is amenable to bedside ultrasonography performed by Intensivists. The investigators hypothesize that measurement of the carotid artery Corrected Flow Time (FTC) in response to a passive leg raise (PLR), which simulates a fluid bolus, can be used to predict fluid responsiveness.

DETAILED DESCRIPTION:
Predicting fluid responsiveness in the Intensive Care Unit (ICU) is a difficult task. Clearly, early aggressive resuscitation in patients with severe sepsis and septic shock improves outcomes. Conversely, overzealous fluid administration is associated with increased mortality in patients with septic shock and acute lung injury. However, recent studies have challenged conventional wisdom that clinical exam, central venous pressure (CVP), or pulmonary artery occlusion pressure (PAOP) are able to predict volume status or fluid responsiveness.

Only approximately 50% of ICU patients have been shown to respond to volume expansion in studies designed to examine fluid responsiveness.9 Ideally, Intensivists would have access to a cheap, reliable, continuously operating, non-invasive, and user friendly device so that fluid could be administered until their patient is no longer fluid responsive. Stroke volume could be maximized via the Frank-Starling relationship and over resuscitation with its potential deleterious effects could be avoided. Although measurement of thermodilution cardiac output by the Pulmonary Artery Catheter (PAC) is considered the "gold standard" by which new devices are validated, it has a waning role in modern ICUs. Existing technologies such as Esophageal Doppler, Transpulmonary Indicator Dilution, and Arterial-Pressure-Waveform-Derived methods, while not as invasive as a PAC, are still invasive procedures. Echocardiography is an excellent tool, however assessing for fluid responsiveness requires advanced training beyond a qualitative approach and it can be difficult to obtain optimal windows in critically ill patients. Thus, current methods for assessment of fluid responsiveness are suboptimal.

The use of Carotid Doppler to determine volume responsiveness has recently been proposed. Remarkably, the authors found that an increase in carotid blood flow of 20% predicted fluid responsiveness with a sensitivity of 94% and specificity of 86%. This appears to be an attractive option, with the caveats that not all point of care ultrasound machines currently available have the software capability to calculate carotid artery velocity time integral (VTI) and this method was validated using Bioreactance, the reliability of which has been recently questioned. A more simple method of evaluating the carotid artery for fluid responsiveness, the Carotid Flow Time, was recently discussed on a popular ultrasound podcast, but has not yet been validated in a clinical study.

The Carotid Artery Corrected Flow Time (FTC) concept is not new. In fact, it has been well studied as a marker of preload and afterload with Transesophageal Doppler (TED). TED monitors display a wave form of the velocity versus time similar to the image one might obtain doing pulsed wave Doppler (PWD) of the carotid artery. With TED, the waveform has a triangular appearance. The apex of the triangle represents peak velocity, which along with mean acceleration reflects cardiac contractility. The area under the systolic portion of the curve is equal to stroke distance, and when multiplied by the cross sectional area of the descending aorta this value can be used to estimate cardiac output predicated on the assumption that the descending aorta receives 70% of cardiac output. The investigators are interested in the base of the triangle representing systolic ejection time. When corrected for heart rate by dividing by the square root of cardiac cycle time we have the FTC. The FTC would be expected to increase with enhanced preload or reduction in afterload; conversely it should decrease with a reduction in preload or increase in afterload. One study performed in 20 neurosurgical patients with TED showed that the FTC was able to predict fluid responsiveness when used as a static measure with a cutoff of 357 ms prior to loading with 7 ml/kg of hydroxyethyl starch solution. The area under the receiver operating curve (ROC) was 0.944.

The investigators believe that the concept of FTC as a marker of preload can be combined conveniently with PWD of the carotid artery and a passive leg raising maneuver (PLR) to estimate fluid responsiveness in critically ill patients. The method is very attractive due to the ease of access to the carotid artery, reproducibility, low cost, and since the FTC is a measurement of time (not velocity), the angle of insonation should be inconsequential, making the exam technically easier to perform compared to carotid artery VTI. This can be compared to a 10% increase in SVI following a PLR demonstrated by the Flotrac/Vigileo being considered the "gold standard". While the absolute values of cardiac output obtained with the Flotrac/Vigileo when compared with the PAC are debatable, the ability of the device to track changes in cardiac output/stroke volume in response to changes in preload and PLR have been shown to be accurate.16-19 A meta-analysis published by Cavallaro and colleagues showed that PLR induced changes in cardiac output were able to predict fluid responsiveness with a sensitivity and specificity of 89.4% and 91.4% with a pooled area under the ROC value of 0.95 regardless of ventilation mode, underlying cardiac rhythm, and technique of measurement. Thus, an increase in SVI > 10% with PLR detected by a Flotrac/Vigileo monitor without the need for a fluid bolus, should be sufficient to determine whether PLR induced changes in carotid FTC are able to detect fluid responsiveness.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older,
* admitted to ICU and already have an arterial line and Flotrac/Vigileo monitor in place ordered by primary team as part of their clinical standard practice.

Exclusion Criteria:

* Not in sinus rhythm,
* clinically suspected or known intraabdominal hypertension,
* lower extremity amputee,
* femoral arterial line,
* poor or unreliable arterial line waveform,
* history of carotid endarterectomy in the artery being measured,
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2014-06; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Fluid Responsiveness | 3 minutes
  Passive leg raise induced increase in stroke volume of 10% on vigileo monitor

CONTACTS AND LOCATIONS:
Locations (1):
- University of Louisville, Louisville, Kentucky, United States